CLINICAL TRIAL: NCT01583049
Title: Observational Post Authorisation Safety Study to Describe the Safety Profile of the Diphtheria, Tetanus, Acellular Pertussis Combination Vaccine, Reduced Antigen Content (Triaxis) as a 5th Dose in 4-6 Year Old Spanish Children
Brief Title: Post Authorisation Safety Study of Triaxis as a 5th Dose in 4-6 Year Old Spanish Children
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: CVX01E
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Diphtheria, Tetanus and Pertussis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary objective: This is a descriptive study and the primary objective is to determine the incidence of injection site and systemic adverse events after Triaxis administration as a 5th dose of tetanus, diphtheria and acellular pertussis vaccine in 4-6 year old children

ELIGIBILITY:
Inclusion Criteria:

* Aged 4 to 6 years on the day of enrolment.
* Have received, on the day of enrolment, immunisation with Triaxis as a 5th dose for diphtheria, tetanus, pertussis vaccination in routine practice in accordance with the Spanish version of the EU SmPC and the Spanish immunisation recommendations.
* Have received a complete course of immunisation with diphtheria, tetanus and pertussis (4 doses).
* Participant and participant´s parent/legal representative are able to comply with all study procedures.
* Written informed consent obtained from at least one parent/legal representative of the participant before the participant is enrolled in the study

Exclusion Criteria:

* Have been previously vaccinated with a 5th dose of tetanus, diphtheria and pertussis.
* Presence of a contra-indication or cautions to vaccination in accordance with the Spanish version of the EU SmPC:

  1. Hypersensitivity to vaccines of diphtheria, tetanus or pertussis, any component of the vaccine and any residual component of the manufacturing process such as formaldehyde and glutaraldehyde that may be present in trace amounts.
  2. Encephalopathy of unknown origin within 7 days after a prior immunisation with a vaccine against pertussis.
  3. Progressive neurological disorder, uncontrolled epilepsy, progressive encephalopathy if no treatment has been established and the condition is not stable.
  4. Acute severe febrile illness or acute infection.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between 4-6 years of age who attend the investigator's office to receive a 5th dose of tetanus, diphtheria and pertussis Triaxis vaccine as part of the routine vaccination schedule, as described in the Spanish version of the EU SmPC and local vaccination calendar
Sampling Method: Non-Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
All Injection Site and Systemic Adverse Events | 30 days following vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (22):
- Spain (22):
  - Centre 11, Almería
  - Centre 12, Almería
  - Centre 13, Almería
  - Centre 14, Almería
  - Centre 15, Almería
  - Centre 16, Almería
  - Centre 17, Almería
  - Centre 18, Almería
  - Centre 19, Almería
  - Centre 20, Almería
  - Centre 21, Almería
  - Centre 22, Almería
  - Centre 10, Madrid
  - Centre 1, Madrid
  - Centre 2, Madrid
  - Centre 3, Madrid
  - Centre 4, Madrid
  - Centre 5, Madrid
  - Centre 6, Madrid
  - Centre 7, Madrid
  - Centre 8, Madrid
  - Centre 9, Madrid